CLINICAL TRIAL: NCT06127550
Title: Effect of Non-invasive Vagus Nerve Stimulation on Letter Learning in Dyslexia
Brief Title: taVNS for Letter Learning in Dyslexia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Waiting on funding to support study
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB202301883
Record Dates: First submitted 2023-10-27; First posted 2023-11-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-02

CONDITIONS: Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either active stimulation or sham stimulation groups.
Who Masked: Participant
Masking Description: All participants will be told they are receiving active stimulation at a custom current level that may or may not be detectable to them. Half of the participants (randomly assigned) will not receive stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active taVNS (Experimental): Participants will receive custom current at 5 Hz to the left auricular branch of the vagus nerve while learning new letter-sound relationships.
  Interventions: Device: active taVNS
- Sham taVNS (Sham Comparator): Participants will undergo current thresholding but device will be turned off without their knowledge during the training.
  Interventions: Device: sham taVNS

INTERVENTIONS:
Device: active taVNS — low level stimulation to the auricular branch of the vagus nerve
  Arms: Active taVNS
Device: sham taVNS — device placed with no current administered
  Arms: Sham taVNS

SUMMARY:
This is a pilot study to establish feasibility of transcutaneous auricular vagus nerve stimulation (taVNS) for improving letter-learning in adolescents with dyslexia. The main goals of the study are to 1) evaluate whether children in this age range will tolerate low level stimulation over the course of multiple sessions, 2) determine whether low level taVNS improves novel letter learning in dyslexia, and 3) evaluate the effect of low level taVNS on the brain's response to letters. Participants will complete fMRI before training, immediately after training, and a few weeks after training ends. Training will consist of six 30-minute lessons during which participants will learn novel letter-sound relationships while receiving either active or sham taVNS. Researchers will compare stimulation conditions to determine effect of this device on learning and neural plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Normal non-verbal IQ
* Reading scores above 90 on four single word reading measures (typical reader) OR reading scores below 90 on two or more single word reading measures (dyslexia) with or without ADHD

Exclusion Criteria:

* Neurological diagnoses (e.g., autism, epilepsy, etc.)
* Medications other than those prescribed for ADHD
* Nonverbal IQ below 80

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 4 weeks
  Frequency and severity of adverse events will be monitored and evaluated for severity and impact on attrition.
Compliance | 4 weeks
  Percentage of the population that remains engaged in the study and completes all stimulation sessions.

SECONDARY OUTCOMES:
Letter ID | 6 weeks
  Percent correct of learned letter-sound relationships
Decoding | 6 weeks
  Percent correct of pseudowords read in 45 seconds
Automaticity | 6 weeks
  This measure is based on a standardized measure for rapid letter naming in English (CTOPP-Rapid Automatized Naming) in which the participant is shown a grid of many letters in Hebrew and are asked to read the grid as quickly and accurately as possible while being timed.

OTHER OUTCOMES:
fMRI | 6 weeks
  Strength of the brain's response to learned letters in the visual word form area

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States